CLINICAL TRIAL: NCT00742859
Title: A Phase 2, Randomized, Parallel Group, Dose-Finding, Multicenter, Multinational Study of the Safety, Tolerability and Pilot Efficacy of Three Blinded Doses of the Oral Factor Xa Inhibitor Betrixaban Compared With Open-Label Dose-Adjusted Warfarin in Patients With Non-Valvular Atrial Fibrillation (EXPLORE Xa)
Brief Title: Phase 2 Study of the Safety, Tolerability and Pilot Efficacy of Oral Factor Xa Inhibitor Betrixaban Compared to Warfarin
Acronym: EXPLORE-Xa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-015
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Betrixaban; Factor Xa inhibitor; Warfarin
MeSH Terms: conditions — Atrial Fibrillation | interventions — betrixaban; Warfarin; Acenocoumarol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1: Betrixaban (Experimental): Betrixaban, 40 mg, orally, once daily for at least 3 months.
  Interventions: Drug: betrixaban
- Arm 2: Betrixaban (Experimental): Betrixaban, 60 mg, orally, once daily for at least 3 months
  Interventions: Drug: betrixaban
- Arm 3: Betrixaban (Experimental): Betrixaban, 80 mg, orally, once daily for at least 3 months
  Interventions: Drug: betrixaban
- Arm 4: Warfarin (Active Comparator): Warfarin will be prescribed by investigators according to the standard of care.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: betrixaban — orally, once daily for at least 3 months
  Arms: Arm 1: Betrixaban; Arm 2: Betrixaban; Arm 3: Betrixaban
Drug: Warfarin — Warfarin will be prescribed by the investigator according to the standard of care.
  Other Names: Coumadin; Acenocoumarol
  Arms: Arm 4: Warfarin

SUMMARY:
Prevention of stroke in patients with atrial fibrillation (AF). Hypothesis: In patients with non-valvular AF, orally administered betrixaban will provide similar or better efficacy and safety than warfarin and it will offer the advantage of not requiring dose adjustments due to international normalized ratios (INRs) outside the target range of 2.0 to 3.0 and a more consistent level of anticoagulation over time.

DETAILED DESCRIPTION:
To assess the safety and tolerability of betrixaban at doses of 40 mg, 60 mg and 80 mg given orally once a day for at least 3 months compared to dose-adjusted warfarin in patients with non-valvular atrial fibrillation (AF).

This is a Phase 2, exploratory, randomized, parallel group, multicenter, active comparator, dose finding study of patients with documented non-valvular AF. Patients will be randomized (1:1:1:1) to 1 of 4 treatment groups (approximately 125 patients per group) using an interactive voice response system (IVRS). A dynamic randomization will be used to balance patients by country, concurrent aspirin use (yes or no) and antecedent warfarin (yes or no). The study will be open label for randomization to warfarin versus betrixaban, but the three daily doses of betrixaban, 40 mg, 60 mg or 80 mg, will be double-blind (identical capsules for all three dose levels). The warfarin-treated patients will be managed according to each center's usual clinical routine with INR monitoring and dose-adjustments in order to maintain a target INR of 2.0 to 3.0 at maximum intervals of four weeks. No loading doses or dose titrations will be used for betrixaban. The betrixaban dose should be ingested in the evening (e.g. at bedtime), preferably at least 2 hours after the evening meal. Note: acenocumerol may be substituted for warfarin as indicated by local practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥18 years.
* If the patient is a woman, she must be without reproductive potential (i.e., postmenopausal for ≥2 years or after hysterectomy).
* AF at the time of enrollment (randomization) or documented within the last year by Holter, ECG, rhythm strip, pacemaker or other intracardiac recording, resulting in an indication for anticoagulation with warfarin, acenocumerol, phenprocoumon, or other Vitamin K antagonist in the opinion of the treating physician.
* One or more of the following risk factor(s) for stroke:

  1. Age 75 years or older.
  2. Prior stroke, TIA or systemic (i.e., central nervous system) embolus at least 30 days remote from the time of screening.
  3. Symptomatic congestive heart failure within 3 months echocardiography, radionuclide study or contrast angiography.
  4. Hypertension requiring pharmacological treatment.
  5. Diabetes.
  6. Age of 55 years or older and previous coronary artery disease or known peripheral artery disease.

Exclusion Criteria:

* Body weight less than 40 kg (88 lbs).
* Need for either hemodialysis or peritoneal dialysis (or likely to require it within one year).
* AF due to reversible causes (e.g., thyrotoxicosis, pericarditis, cardiac surgery, pulmonary embolism).
* Mechanical prosthetic valve (bioprosthetic valve is allowed) or valvular disease likely to be operated on within one year.
* History (including family history) or symptoms of a congenital or acquired bleeding disorder or vascular malformation; or a history of intracranial, retroperitoneal, or intraocular bleeding within the last 6 months; or is felt to be at high risk for bleeding for other reasons including from significant liver disease. This also includes gastrointestinal bleeding within 90 days before randomization or endoscopically verified ulcer disease within 30 days of screening.
* Conditions other than AF that require chronic anticoagulation (e.g. prosthetic mechanical heart valve).
* Persistent, uncontrolled hypertension (SBP >160 mm Hg on repeated measurements).
* Active infective endocarditis.
* Scheduled major surgery.
* Planned pulmonary vein ablation or surgical procedure for cure of AF or flutter.
* Recent ischemic stroke, systemic embolic event or acute coronary syndrome within 30 days.
* Severe co-morbid condition with life expectancy of ≤1 year.
* Previous known history of genetic coagulopathy (e.g., Factor V Leiden, Protein C Deficiency, Protein S Deficiency, Antiphospholipid Syndrome, etc.).
* Evidence at Screening of:

  1. Platelet count <100,000/mm3.
  2. Serum alanine aminotransferase (ALT) or aspirate aminotransferase (AST) >2 times upper limit of normal (ULN).
  3. A history (including family history) of "Long QT Syndrome".
* Aspirin >162 mg daily.
* Use of verapamil (pending the availability of a drug interaction study with betrixaban).
* Active alcohol or drug abuse, or psychosocial reasons that make study participation impractical.
* Use of an investigational drug or device within the past 30 days.
* Inability to comply with INR monitoring or other protocol-related activities.
* Unable to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Connolly, MD, FRCP, Study Chair — Population Health Research Institute, McMaster University; Rafael Diaz, MD, Study Director — Instituto Cardiovascular de Rosario, Argentina; Paul Dorian, MD, Study Director — University of Toronto, Canada; Michael Ezekowitz, MD, PhD,, Study Director — Lankenau Institute for Medical Research and The Heart Center, United States; Stefan H. Hohnloser, MD, Study Director — Johann Wolgang Goethe University, Frankfurt, Germany
Locations (21):
- United States (19):
  - Portola Investigational Site, Anaheim, California
  - Portola Investigational Site, Colorado Springs, Colorado
  - Portola Investigational Site, Melbourne, Florida
  - Portola Investigational Site, Miami, Florida
  - Portola Investigational Site, Ormond Beach, Florida
  - Portola Investigational Site, Pensacola, Florida
  - Portola Investigational Site, Port Charlotte, Florida
  - Portola Investigational Site, Aurora, Illinois
  - Portola Investigational Site, Auburn, Maine
  - Portola Investigational Site, Columbia, Maryland
  - Portola Investigational Site, Salisbury, Maryland
  - Portola Investigational Site, Towson, Maryland
  - Portola Investigational Site, Tupelo, Mississippi
  - Portola Investigational Site, St Louis, Missouri
  - Portola Investigational Site, Poughkeepsie, New York
  - Portola Investigational Site, Hillsboro, Oregon
  - Portola Investigational Site, Wynnewood, Pennsylvania
  - Portola Investigational Site, Rapid City, South Dakota
  - Portola Investigational Site, Norfolk, Virginia
- Canada (2):
  - Portola Investigational Site, Longueuil, Quebec
  - Portola Investigational Site, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 31 October 2008 and 05 November 2009, 508 patients were enrolled by 35 study centers in 3 countries (USA, Canada, Germany). Patients were randomized to 1 of 4 treatment groups (1:1:1:1 allocation). The study was open-label for warfarin, while the 3 daily doses of betrixaban (40, 60, or 80 mg) were double-blinded.
Pre-assignment Details: 561 patients were screened for study participation. Of these patients, 508 were randomized, all of whom received at least 1 dose of study drug.
Groups:
- Betrixaban 40 mg: Betrixaban 40 mg once daily for at least 3 months and no longer than approximately 11 months
- Betrixaban 60 mg: Betrixaban 60 mg once daily for at least 3 months and no longer than approximately 11 months
- Betrixaban 80 mg: Betrixaban 80 mg once daily for at least 3 months and no longer than approximately 11 months
- Warfarin: Dose-adjusted warfarin to maintain an INR of 2.0 to 3.0 with INR measured at maximum intervals of 4 weeks. Treatment duration was at least 3 months and no longer than approximately 11 months
Period: Overall Study
Arm/Group | Betrixaban 40 mg | Betrixaban 60 mg | Betrixaban 80 mg | Warfarin
Started | 127 | 127 | 127 | 127
Completed | 116 | 115 | 116 | 119
Not Completed | 11 | 12 | 11 | 8
Not completed — Adverse Event | 5 | 6 | 3 | 1
Not completed — Death | 1 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 4 | 1
Not completed — Endpoint | 0 | 1 | 1 | 2
Not completed — Amendment 2 patient off study drug >4wks | 0 | 1 | 1 | 0
Not completed — Sponsor req visit schedule noncompliance | 0 | 0 | 0 | 1
Not completed — Sponsor request patient out of town | 0 | 0 | 1 | 1
Not completed — Site error | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients who took at least 1 dose of study medication after randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Betrixaban 40 mg | Betrixaban 60 mg | Betrixaban 80 mg | Warfarin | Total
Number analyzed (Participants) | 127 | 127 | 127 | 127 | 508
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (8.50) | 73.8 (8.35) | 72.0 (7.65) | 72.7 (8.75) | 73.0 (8.32)
Age, Customized [Number; unit: Count of Participants]
  <75 years | 64 | 61 | 76 | 67 | 268
  >=75 years | 63 | 66 | 51 | 60 | 240
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 38 | 38 | 170
  Male | 79 | 81 | 89 | 89 | 338

OUTCOME MEASURES:

1. Primary Outcome: Exposure-adjusted Incidence Rate of Major or Clinically Relevant Non-major Bleeding Episode
Description: The primary endpoint is the time to the first occurrence of major or clinically relevant non-major bleeding. This was presented as the exposure adjusted incidence rate which was calculated as number of subjects experiencing the event divided by total person years across all subjects, where if a patient experiencing the event, year was from first dose date to the first occurrence of the event, and to last study date if not. The confidence interval was calculated via the exact Poisson distribution.
Time Frame: A maximum of 1 year
Population: All randomized patients who took at least 1 dose of study medication after randomization.
Measure: Number (95% Confidence Interval); unit: Number of Patients per 100 Patient years
Arm/Group | Betrixaban 40 mg | Betrixaban 60 mg | Betrixaban 80 mg | Warfarin
Number analyzed (Participants) | 127 | 127 | 127 | 127
Number of Patients per 100 Patient years | 2.02 [0.05 to 11.3] | 10.1 [3.28 to 23.6] | 10.5 [3.41 to 24.5] | 14.6 [5.85 to 30.0]
Statistical Analysis 1: Comparison: Betrixaban 40 mg vs Warfarin; Betrixaban 40mg compared to Warfarin; Test type: Other; p = 0.035, Log Rank; Hazard Ratio (HR) = 0.14, 95% CI 2-sided [0.017 to 1.14]
Statistical Analysis 2: Comparison: Betrixaban 60 mg vs Warfarin; Betrixaban 60mg compared to Warfarin; Test type: Other; p = 0.546, Log Rank; Hazard Ratio (HR) = 0.711, 95% CI 2-sided [0.225 to 2.24]
Statistical Analysis 3: Comparison: Betrixaban 80 mg vs Warfarin; Betrixaban 80mg compared to Warfarin; Test type: Other; p = 0.712, Log Rank; Hazard Ratio (HR) = 0.755, 95% CI 2-sided [0.239 to 2.39]

2. Secondary Outcome: Exposure-adjusted Incidence Rate of Any Bleeding (Major, Clinically Relevant Non-major, or Minimal)
Description: The time to the first occurrence of any bleeding event. This was presented as the exposure adjusted incidence rate which was calculated as number of subjects experiencing the event divided by total person years across all subjects, where if a patient experiencing the event, year was from first dose date to the first occurrence of the event, and to last study date if not. The confidence interval was calculated via the exact Poisson distribution.
Time Frame: A maximum of 1 year
Population: All randomized patients who took at least 1 dose of study medication after randomization.
Measure: Number (95% Confidence Interval); unit: Number of Patients per 100 Patient years
Arm/Group | Betrixaban 40 mg | Betrixaban 60 mg | Betrixaban 80 mg | Warfarin
Number analyzed (Participants) | 127 | 127 | 127 | 127
Number of Patients per 100 Patient years | 50.5 [31.7 to 76.5] | 77.9 [53.3 to 110] | 56.0 [35.9 to 83.4] | 103 [73.6 to 140]
Statistical Analysis 1: Comparison: Betrixaban 40 mg vs Warfarin; Betrixaban 40mg compared to Warfarin; Test type: Other; p = 0.011, Log Rank; Hazard Ratio (HR) = 0.508, 95% CI 2-sided [0.301 to 0.856]
Statistical Analysis 2: Comparison: Betrixaban 60 mg vs Warfarin; Betrixaban 60mg compared to Warfarin; Test type: Other; p = 0.308, Log Rank; Hazard Ratio (HR) = 0.767, 95% CI 2-sided [0.481 to 1.22]
Statistical Analysis 3: Comparison: Betrixaban 80 mg vs Warfarin; Betrixaban 80mg compared to Warfarin; Test type: Other; p = 0.022, Log Rank; Hazard Ratio (HR) = 0.551, 95% CI 2-sided [0.332 to 0.914]

ADVERSE EVENTS:
Time Frame: Maximum of 1 year
Arm/Group | Betrixaban 40 mg | Betrixaban 60 mg | Betrixaban 80 mg | Warfarin
All-Cause Mortality (participants affected / at risk) | 61/127 | 68/127 | 53/127 | 50/127
Serious Adverse Events (participants affected / at risk) | 12/127 | 12/127 | 11/127 | 12/127
Other Adverse Events (participants affected / at risk) | 61/127 | 68/127 | 53/127 | 50/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Betrixaban 40 mg (N=127) | Betrixaban 60 mg (N=127) | Betrixaban 80 mg (N=127) | Warfarin (N=127)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 3
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0 | 0 | 0
Sick Sinus Syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cardiac Neoplasm Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Grand Mal Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Ligament Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arterial Stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Internaional Normalised Ratio Increased (Investigations) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Prostatic Obstruction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Betrixaban 40 mg (N=127) | Betrixaban 60 mg (N=127) | Betrixaban 80 mg (N=127) | Warfarin (N=127)
NAUSEA (Gastrointestinal disorders) | 2 | 5 | 14 | 2
DIARRHOEA (Gastrointestinal disorders) | 4 | 10 | 9 | 1
HEADACHE (Nervous system disorders) | 5 | 6 | 9 | 3
OEDEMA PERIPHERAL (General disorders) | 8 | 10 | 6 | 11
DIZZINESS (Nervous system disorders) | 12 | 9 | 6 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 6 | 6 | 2
VOMITING (Gastrointestinal disorders) | 1 | 2 | 6 | 1
INSOMNIA (Psychiatric disorders) | 2 | 4 | 5 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 5 | 2
FATIGUE (General disorders) | 7 | 5 | 4 | 4
BRONCHITIS (Infections and infestations) | 1 | 2 | 4 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 1 | 4 | 3
INFLUENZA (Infections and infestations) | 2 | 1 | 4 | 1
DYSPEPSIA (Gastrointestinal disorders) | 7 | 0 | 4 | 1
CONSTIPATION (Gastrointestinal disorders) | 9 | 8 | 3 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 3 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 6 | 3 | 4
NASOPHARYNGITIS (Infections and infestations) | 5 | 5 | 3 | 10
RASH (Skin and subcutaneous tissue disorders) | 4 | 3 | 3 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 5 | 2 | 1
CHEST PAIN (General disorders) | 5 | 1 | 2 | 3
URINARY TRACT INFECTION (Infections and infestations) | 3 | 1 | 2 | 4
HYPERTENSION (Vascular disorders) | 3 | 3 | 1 | 4
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 1 | 4
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 | 4 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Due to multiple studies, centers and countries this may vary.